CLINICAL TRIAL: NCT04369859
Title: Obstetric and Perinatal Outcomes of Women With COVID-19: A Prospective Cohort Study
Brief Title: Obstetric and Perinatal Outcomes of Women With COVID-19
Acronym: GROCO
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-18; ID RCB (Other: 2020-A00819-30)
Record Dates: First submitted 2020-04-29; First posted 2020-04-30 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Pregnant Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant women with COVID-19: Pregnant women who have tested positive for COVID-19
  Interventions: Behavioral: Examine the impact of COVID-19 during pregnancy

INTERVENTIONS:
Behavioral: Examine the impact of COVID-19 during pregnancy — clinical data collection

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is currently spreading rapidly around the globe, causing a major public health issue. There is currently very few data about the impact of COVID-19 on pregnancy, and potential in utero infection. This is a prospective observational study of COVID-19 diagnosed pregnant patients. This objective is to examine the impact of COVID-19 during pregnancy on the rates of obstetric and perinatal complications.

DETAILED DESCRIPTION:
Clinical manifestations of COVID-19 can range from a benign upper respiratory tract infection to severe acute respiratory distress syndrome (ARDS), fatal in 1% of cases. However, pregnant women and their fetuses could particularly be vulnerable to the infection, as shown by previous human coronavirus outbreaks (SARS-CoV and MERS-CoV).

Cases will be recruited among all pregnant women aged >18 years old who have tested positive for COVID-19 and are followed in a maternity belonging to the French South Regional Perinatology Network. Voluntary physicians will refer eligible participants to the study-coordinating center at APHM University Hospital. The participants will be followed by phone after having provided an informed consent. Clinical symptoms, laboratory and imaging findings, maternal and perinatal outcomes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Able to give informed consent
* Diagnosed with COVID-19

Exclusion Criteria:

* Patients Refusing to Participate in the Study
* Patients who do not speak French well enough to benefit from clear and intelligible information

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Persons assigned gender female at birth
Study Population: Cases will be recruited among all pregnant women aged >18 years old who have tested positive for COVID-19 and are followed in a maternity belonging to the French South regional perinatology network
Sampling Method: Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-01-15 (Actual)

PRIMARY OUTCOMES:
Compare the complications rates | 12 months
  To compare the complications rates of pregnant women tested positive for the SARS-CoV-2 (study group), with reference rates in a Covid-free population.

SECONDARY OUTCOMES:
Clinical presentation | 12 months
  To record clinical presentation of pregnant participants with COVID-19 by questionnaire and clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, PACA, France

IPD SHARING:
Plan to Share IPD: No